CLINICAL TRIAL: NCT04415424
Title: A Multi-centre Randomised Controlled Trial Evaluating the Efficacy of the Four-component Meningococcal B Vaccine, 4CMenB (Bexsero®), in the Prevention of Neisseria Gonorrhoeae Infection in Gay and Bisexual Men
Brief Title: Efficacy Study of 4CMenB (Bexsero®) to Prevent Gonorrhoea Infection in Gay and Bisexual Men
Acronym: GoGoVax
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Griffith University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HEPP2001; APP1182443 (Other Grant/Funding Number: National Health and Medical Research Council, Australia)
Record Dates: First submitted 2020-05-19; First posted 2020-06-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Neisseria Gonorrheae Infection
MeSH Terms: conditions — Gonorrhea | interventions — 4CMenB vaccine

STUDY DESIGN:
Intervention Model Description: Randomised 1:1 to receive 4CMenB vaccine or a matching placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, their study clinicians and study researchers assessing the outcomes will be blinded to the treatment arm (4CMenB vaccine or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm A - 4CMenB vaccine (Experimental): 4CMenB vaccine will be administered as an intramuscular injection in 0.5 ml single-dose pre-filled syringe in two doses with 3-month apart (at Baseline and Month 3 visit).
  Interventions: Biological: 4CMenB vaccine
- Treatment arm B - placebo (Placebo Comparator): Placebo will be administered as an intramuscular injection in 0.5 ml single dose pre-filled syringe in two doses with 3-month apart (at Baseline and Month 3 visit).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 4CMenB vaccine — A four-component meningococcal B vaccine
  Other Names: Bexsero®
  Arms: Treatment arm A - 4CMenB vaccine
Other: Placebo — 0.5 ml of 150 mmol sodium chloride (0.9% saline solution)
  Arms: Treatment arm B - placebo

SUMMARY:
This is a Phase 3, double-blinded, randomised placebo-controlled, multi-centred trial evaluating the efficacy of the four-component meningococcal B vaccine, 4CMenB (Bexsero®), in the prevention of Neisseria gonorrhoeae infection.The targeted population is 18-50 years-old men (cis and trans), trans women and non-binary people who have sex with men (hereafter referred to as Gay Bisexual Men+ [GBM+], either HIV-negative and taking pre-exposure prophylaxis [PrEP], or HIV-positive with undetectable viral load <200copies/ml and a cluster of differentiation 4 [CD4] count >350 cells/cmm) who have high N. gonorrhoeae incidence and are recommended by Australian guidelines to have regular, comprehensive sexual health screening. 730 participants will be enrolled and randomised 1:1 and stratified by clinical sites to receive two doses of 4CMenB vaccine or a matching placebo at 0 and 3 months by intramuscular injection. Recruitment is for 12 months and all participants will be follow-up 3-monthly for a period of 2 years. The trial aims to evaluate the efficacy of 4CMenB in the prevention of N. gonorrhoeae infection.

DETAILED DESCRIPTION:
This is a Phase 3, double-blinded, randomised placebo-controlled, multi-centred trial evaluating the efficacy of the four-component meningococcal B vaccine, 4CMenB (Bexsero®), in the prevention of Neisseria gonorrhoeae infection.The target population for this trial is GBM+, either HIV-negative and on PrEP or HIV-positive, who had a diagnosis of gonorrhoea or infectious syphilis in the last 18 months (a key characteristic associated with greater gonorrhoea risk). This population has the highest known gonococcal incidence and are recommended under Australian guidelines to attend clinics 3-monthly for comprehensive sexual health screening, including Nuclei acid amplification test (NAAT)-based screening of urine, and pharyngeal and anal specimens for N. gonorrhoeae infection. 730 participants will be enrolled and randomised 1:1 and stratified by clinical sites to receive two doses of 4CMenB vaccine or a matching placebo at 0 and 3 months by intramuscular injection. Recruitment will occur over a 12-month period and all participants will be followed up 3-monthly over a period of 2 years. Participants, their study clinicians and study researchers assessing the outcomes will be blinded to the treatment arm (vaccine or placebo). Participants will be required to attend approximately 10 study visits. Participants may attend additional visits if they have been diagnosed with gonorrhoea infection (symptomatic or asymptomatic) or have a postitive gonorrhoea NAAT test when they return for test of cure. Potentially eligible individuals will be screened within 14 days of baseline (the visit when the first dose of study treatment is administered). Randomisation can be conducted any time between screening and baseline. Screening, randomisation and baseline can occur on the same day if the required HIV result(s) and drug kit (containing 4CMenB or placebo) are available for a participant in the clinic. At screening, study clinicians will conduct the informed consent process with a participant and the informed consent will be signed by both the study clinician and the participant. Eligibility criteria will be checked and a review of medical history (including vaccination history for 4CMenB, prior known meningococcal disease, recent history of sexually transmitted infections [STIs], history of taking PrEP [for HIV negative individuals] as well as antibiotic use in the last 3 months) will be conducted. Routine blood, urine and swabs will be collected, and urine pregnancy test will be performed in participants with child-bearing potential. Symptoms of urethritis, proctitis, epididymitis, and cervicitis/vaginitis will be documented. At randomisation (which can occur anytime within screening an baseline), participants will be randomised to receive either the 4CMenB vaccine or the placebo. At the baseline visit, research blood specimen and an oral mucosal exudate swab for immune responses testing will be collected before the administration of the first dose of the study treatment. A 10-minute study questionnaire will be completed by the participants. Participants will return to their study site 3 months after the first dose of study treatment to receive the second dose. Prior to the treatment administration, urine pregnancy test (in participants with child-bearing potential) will be conducted. Symptoms of urethritis, proctitis, epididymitis, and cervicitis/vaginitis will be documented. History of antibiotic use in the last 3 months will also be collected. If a participant has tested positive for gonorrhoea infection, routinely collected culture isolates and NAAT samples will be stored in a study research laboratory for phenotypic antimicrobial resistance (AMR) testing and genotyping. Routine blood, urine and swabs will also be collected. Adverse events and serious adverse events (SAEs) will be recorded but only SAEs will be entered into the study electronic data capture system, and reported to the Sponsor in real time. Three-monthly visits will be conducted over a period of 2 years. The study aims to evaluate the efficacy of 4CMenB in the prevention of N. gonorrhoeae infection.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 to ≤ 50 years of age
2. Men (cis and trans), trans women and non-binary people who have had sex with at least one man in the last 6 months
3. Diagnosis of gonorrhoea or infectious syphilis in the last 18 months
4. Committed not to take doxycycline as prophylaxis for the duration of the trial
5. Able to understand spoken and written English
6. Willing and likely to comply with the trial procedures for 2 years
7. Agree to be contacted via short message service (SMS)/phone/ email by the study team

AND EITHER

1. HIV-negative (with an HIV negative antibody test within 4 months of screening) and taking HIV PrEP (daily PrEP or on-demand PrEP) within the last 4 months at the time of enrolment or
2. HIV-positive and on an antiviral regimen, with an undetectable virus level of <200 copies/ml and a CD4 count >350 cells/cmm (to optimise the immune response to vaccine) within 12 months of screening

Exclusion Criteria:

1. Have a previous history of vaccination for meningococcal B with 4CMenB
2. Have contraindications to receiving the meningococcal B vaccine which include:

   * Anaphylaxis following a previous dose of any meningococcal vaccine
   * Anaphylaxis following any vaccine component
3. Are participating in biomedical prevention strategies for bacterial STIs (participation in diagnostic or treatment studies is not an exclusion)
4. Are taking long-term (> 4 weeks) antibiotic for prophylaxis or treatment for acne, malaria, syphilis or other bacterial condition(s)
5. Have defects in, or deficiency of, complement components, including factor H, factor D or properdin deficiency
6. Are taking or will receive complement inhibitors such as eculizumab (a monoclonal antibody directed against complement component C5) or ravulizumab
7. Have functional or anatomical asplenia, including sickle cell disease or other haemoglobinopathies, and congenital or acquired asplenia
8. Have had a haematopoietic stem cell transplant
9. Have any major unstable medical condition or therapy that may cause immune compromise (e.g. chemotherapy, radiation, corticosteroids [prednisone >5mg/day] within 14 days prior to screening)
10. Documented allergy to latex and/or kanamycin
11. Have prior known meningococcal disease
12. Positive pregnancy test at screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — High risk men (cis and trans), trans women and non-binary people who have sex with men (hereafter referred to as GBM+)
Enrollment: 650 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
To measure whether the 4CMenB vaccine, when administered in a 2-dose regimen at 0 and 3 months, changes the incidence of the first episode of N. gonorrhoeae. | From Month 4 to Month 24
  Detection of the first instance of N. gonorrhoeae infection in a urine sample or on a swab taken from the urethra, anorectum, oropharynx or vagina, as determined by nucleic acid amplification (NAAT) testing.
To compare the overall incidence of all episodes of N. gonorrhoeae infection diagnosed during the study period between the vaccine and placebo arms. | From Month 4 to Month 24
  To compare the overall incidence of all episodes of N. gonorrhoeae infection diagnosed during the study period between the vaccine and placebo arms, allowing multiple diagnoses of N. gonorrhoeae infection occurred in the same individuals at different time points.

SECONDARY OUTCOMES:
To measure the impact of administration of a 2-dose regimen of 4CMenB vaccine on the incidence of the first episode of symptomatic N. gonorrhoeae infection of the urethra, anorectum or vagina. | From Month 4 to Month 24
  Symptomatic N. gonorrhoeae infection - first instance of the detection of N. gonorrhoeae infection in a urine sample or on a swab taken from the urethra, anorectum or vagina at a study visit when a participant also reports any symptoms at the relevant anatomic site.
To measure the impact of administration of a 2-dose regimen of 4CMenB vaccine on the incidence of the first episode of asymptomatic N. gonorrhoeae infection of the urethra, anorectum, oropharynx or vagina. | From Month 4 to Month 24
  Asymptomatic N. gonorrhoeae infection - first instance of the detection of N. gonorrhoeae infection in a urine sample or on a swab taken from the urethra, anorectum, oropharynx or vagina at a study visit when a participant reports no symptoms at the relevant anatomic site.
To measure the impact of administration of a 2-dose regimen of 4CMenB vaccine on the incidence of first episode of N. gonorrhoeae infection, regardless of symptoms and anatomic sites, by various N. gonorrhoeae strain types (genotype and AMR phenotype). | From Month 4 to Month 24
  Strain specific (by whole genome sequence or antimicrobial resistance phenotype) - first instance of the detection of N. gonorrhoeae infection in a urine sample or on a swab taken from the urethra, anorectum, oropharynx or vagina, at a study visit.

OTHER OUTCOMES:
To evaluate if the N. gonorrhoeae-specific enzyme-linked immunosorbent assay (ELISA) titres increase following 4CMenB vaccination. | From Baseline through to Month 3
  The enzyme-linked immunosorbent assay (ELISA) of serum and oral mucosal transudates post 4CMenB dose 1 and dose 2, relative to baseline.
To evaluate if the N. gonorrhoeae-specific serum bactericidal activity assay titres increase following 4CMenB vaccination. | From Baseline through to Month 3
  The serum bactericidal activity (SBA) titres of serum post 4CMenB dose 1 and dose 2, relative to baseline.
To evaluate if the serum opsonophagocytic killing assay (OPK) titres increase following 4CMenB vaccination. | From Baseline through to Month 3
  The opsonophagocytic killing (OPK) titres of serum post 4CMenB dose 1 and dose 2, relative to baseline.
To evaluate if the N. gonorrhoeae-specific ELISA correlate with reduced N. gonorrhoeae infection. | From Baseline through to Month 24
  The ELISA titres of serum during the study period.
To evaluate if the N. gonorrhoeae-specific titres correlate with reduced N. gonorrhoeae infection. | From Baseline through to Month 24
  The SBA titres of serum during the study period.
To evaluate if the N. gonorrhoeae-specific OPK titres correlate with reduced N. gonorrhoeae infection. | From Baseline through to Month 24
  The OPK titres of serum during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Kate Seib, BSc(Hon),PhD, Study Chair — Institute for Glycomics, Griffith University, Queensland, Australia; Professor Basil Donovan, MBBS, MD, Principal Investigator — The Kirby Institute, University of New South Wales Sydney, Australia; Professor Andrew Grulich, MBBS, PhD, Principal Investigator — The Kirby Institute, University of New South Wales Sydney, Australia
Locations (7):
- Australia (7):
  - Western Sydney Sexual Health Centre, Parramatta, New South Wales
  - Sydney Sexual Health Centre, Sydney, New South Wales
  - Taylor Square Private Clinic, Sydney, New South Wales
  - RPA Sexual Health, Sydney, New South Wales
  - Gold Coast Sexual Health Service, Southport, Queensland
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Prahran Market Clinic, Melbourne, Victoria

REFERENCES:
- [Derived] Seib KL, Donovan B, Thng C, Lewis DA, McNulty A, Fairley CK, Yeung B, Jin F, Fraser D, Bavinton BR, Law M, Chen MY, Chow EPF, Whiley DM, Mackie B, Jennings MP, Jennison AV, Lahra MM, Grulich AE. Multicentre double-blind randomised placebo-controlled trial evaluating the efficacy of the meningococcal B vaccine, 4CMenB (Bexsero), against Neisseria gonorrhoeae infection in men who have sex with men: the GoGoVax study protocol. BMJ Open. 2024 Apr 16;14(4):e081675. doi: 10.1136/bmjopen-2023-081675. PMID 38626958